CLINICAL TRIAL: NCT03336736
Title: The Role of Non-pharmacological Rehabilitation Within Pulmonary Sarcoidosis: The Role of Physical Activity and Diet Within Pulmonary Sarcoidosis
Brief Title: The Role of Physical Activity and Diet Within Pulmonary Sarcoidosis
Status: Completed | Type: Observational
Sponsor: Kingston University (Other)
Responsible Party: Principal Investigator, Hannah Moir, Principal Investigator- Senior Lecturer in Health & Exercise Prescription, Kingston University
Other Study IDs: KingstonUSport
Record Dates: First submitted 2017-07-19; First posted 2017-11-08 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Sarcoidosis; Sarcoidosis, Pulmonary; ILD; Interstitial Lung Disease
Keywords: Physical Activity; Diet; Exercise; Sarcoidosis; Pulmonary sarcoidosis; Lung Function; Fitness; Strength; Endurance
MeSH Terms: conditions — Sarcoidosis; Sarcoidosis, Pulmonary; Lung Diseases, Interstitial; Motor Activity | interventions — Exercise

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pulmonary Sarcoidosis: Self-reported and self-referred self-reported medically diagnosed pulmonary sarcoidosis.
  Exercise capacity and function will be assessed.
  Interventions: Diagnostic Test: Exercise
- Control: Healthy age-matched control group with no known lung disease. Exercise capacity and function will be assessed.
  Interventions: Diagnostic Test: Exercise

INTERVENTIONS:
Diagnostic Test: Exercise — The study design will be a prospective cross-sectional observational project, with no intervention.
  Data on a participant's physical activity levels, physical fitness and quality of life will be collected using physical testing and questionnaires.

SUMMARY:
This project focuses on the sub-group population with pulmonary sarcoidosis - a condition that causes red swollen tissue called granulomas to develop in organs such as the lungs. The condition is associated to symptoms of shortness of breath and a persistent dry cough. The aim of the research is to investigate the role of physical activity, exercise and diet within pulmonary sarcoidosis-related outcomes. Exercise has the potential to improve symptoms of pulmonary sarcoidosis including fatigue, dyspnoea, quality of life (QOL) and exercise tolerance. The use of exercise in symptomatic patients is supported by current evidence but is limited and requires further understanding, given the unique nature of the condition, in terms of physical and psychological outcomes. Specific dietary and exercise recommendations are limited by the lack of evidence for specific modifications such as the type(s), intensities, frequency and duration.

The study will involve completion of validated questionnaires including quality of life (QOL; Sarcoidosis Health Questionnaire (SHQ) (see appendix III), the SHQ comprises of 29-item, 7 point Likert scale questionnaire and fatigue (Fatigue Assessment Scale; FAS (see appendix IV) and will require participants to attend two visits to the Kingston University, Human Performance Lab at Penrhyn Rd campus, this is to ensure reliability and validity for the data collected. The visits will consist of a range of physical tests including lung function, a six-minute walk test and muscle strength tests. The primary aim of the study is to ascertain the physical activity patterns in those with pulmonary sarcoidosis with regards to perceived physical activity, measured using the the International Physical Activity Questionnaires (IPAQ) (appendix V), which comprises of 27 items across five activity domains and actual physical activity ,measured by tri-axial accelerometry, fatigue assessment scale (appendix IV). The secondary aim of the study is to understand the effect of pulmonary sarcoidosis in relation to muscle strength and exercise capacity against physical activity, lung function and oxygen saturation and how these differ from healthy normative values.

Participants will be asked to read the participant information and declare consent before starting the study. Only the researcher and supervisors of the study will have access to the raw data. Anonymity will be kept all times.

DETAILED DESCRIPTION:
This is a prospective cross-sectional observational project, with no intervention. All data will be self-reported and self-referred for voluntary participation. The participant information sheet and consent form will be provided in advance following interest of participation from the volunteers via email. In addition, on voluntary consent and approval of participation, the participant's general practitioner (GP) or consultant will be informed of their involvement in the study. Participants will be recruited via online forums, social media sources and via the newsletters /communication from Sarcoidosis organisations and Charities (e.g. The Sarcoidosis Charity; Sarcoidosis UK, Breathing Matters). Travel cost reimbursement will be offered to all participants who attend lab visits.

During visit one, participants will sign informed consent forms and have any questions answered before continuing. Baseline characteristics such as anthropometric data (stature, mass, heart rate (HR), blood pressure, age, BMI, fat% (Bodpod, Cosmed/ Bioelectric Impedance Analysis (BIA), Tanita) will be collected. Following this, participants will conduct a lung function test via computer spirometry (Oxycon Pro, VIASYS GmbH, Eric Jaeger, Hoechberg, Germany) and their predicted results will be corrected for ethnicity, allowing an accurate percentage of lung function to be recorded (Caucasian results remain the same, whilst Black-Caribbean are decreased by 13%). Participants will then conduct muscle strength testing of key muscle groups using an isokinetic dynamometer (Biodex System 4,Biodex Corporation, NY, USA); tests include: elbow flexor muscle strength (EFMS), quadriceps peak torque (QPT) and hamstring peak torque (HPT), in addition to this handgrip strength will also be assessed via handgrip digital dynamometer (Accord Medical Products; appendix XII). A minimum rest period of 20 minutes will follow based on exercise-based pulmonary rehabilitation research. Heart rate (bpm) will be checked at the end of this period and in two minute intervals until HR returns to baseline as per American College of Sport Medicine (ACSM) guidelines. Physical testing will not take place until this return to baseline. Following this rest period, participants will conduct a six-minute walk test (6MWT; appendix VIII). During the test participants will be measured for Borg rate of perceived exertion (appendix IX) and Borg Dyspnoea (appendix X) at 2 minute intervals and at completion of the test. Oxygen saturation (SO2) levels of participants will be recorded during the 6MWT via a portable pulse oximeter. Once the 6MWT has been completed participants will complete three questionnaires, the fatigue assessment scale (FAS; appendix IV), international physical activity questionnaire (IPAQ; appendix V) and Sarcoidosis Health Questionnaire (SHQ; Cox et al., 2003; appendix III). Before leaving, participants will be given a tri-axial accelerometer to wear on their hip (GT3X+ accelerometer, Actigraph) via a belt clip, which will be used to measure the participant's physical activity (PA) for seven days, to establish habitual physical activity levels and compare against the results of the IPAQ.

During the second lab visit, participants will return their accelerometers and following the same pattern of testing as the first visit, excluding the questionnaires (SHQ, FAS & IPAQ) and anthropometric information. The order of testing will follow ACSM guidelines therefore strength and aerobic/anaerobic capacity will be first. Alongside this, age-matched healthy participants with no known interstitial lung disease (ILD) or other condition linked to reduced physical activity will used as a comparison between sarcoidosis and healthy normative values.

Procedural details:

* Six Minute Walk Test: Performed along a straight flat 30 metre course indoors, participants walk at their own pace for 6 minutes. No warm-up is required however participants rest in the seated 10 minutes before the test in accordance with American Thoracic Society guidelines.
* International Physical Activity Questionnaire (IPAQ): IPAQ comprises of 27 items across five activity domains asked independently.
* Fatigue Assessment Scale (FAS): - FAS is a 10-item questionnaire with a 5-point Likert scale, it is split into 5 physical fatigue and 5 mental fatigue questions.
* Sarcoidosis Health Questionnaire (SHQ): SHQ is a 29-item questionnaire with a 7-point Likert scale.
* Borg rate of perceived exertion and Borg Dyspnoea: The Borg rate of perceived exertion scale (Borg RPE) allows participants to express how exerted they feel via a numbered scale, modified Borg Dyspnoea scale (Borg DS) allows participants to express their shortness of breath.
* Distance Saturation Product (DSP): DSP is calculated by multiplying the distance a participant walks against their lowest oxygen saturation (Sp02) recorded during the 6MWT.
* Oxygen saturation levels (SpO2): Oxygen saturation levels of participants will be recorded during the 6MWT via a portable pulse oximeter, the device will be fitted to the participant's finger and checked every 30 seconds throughout.
* Isokinetic Dynamometer: A Biodex system will be utilized to look at dominant upper and lower limb strength via elbow flexor muscle strength (EFMS), quadriceps peak torque (QPT) and hamstring peak torque (HPT) tests, with rest periods of 60 seconds between repeated tests as per previous research findings.
* Hand Dynamometer: Utilised to measure hand grip strength following ACSM guidelines.
* Tri-axial Accelerometer: Participants will keep this on their persons throughout the time between their lab visits to measure real world physical activity for seven days.

ELIGIBILITY:
Inclusion Criteria:

* Patients with known Sarcoidosis according to ATS/ERS/ WASOG criteria statement
* Written informed consent is obtained.
* Access to a computer with Internet

Exclusion Criteria:

* Contraindications to (not able to perform) physical tests or exercise testing - e.g. unstable cardiovascular disease, oncological, cardiac, neurological or orthopaedic history making them unable to participate screened by a sub-maximal fitness screening form (appendix ).
* An injury in the past 6 months that inhibits ability to perform exercise testing by a sub-maximal fitness screening form (appendix).
* Patients with a concurrent and predominant diagnosis of another significant respiratory disorder (for example: asthma, chronic obstructive pulmonary disease (COPD), cystic fibrosis, or lung cancer) by a sub-maximal fitness screening form (appendix).
* Pregnancy
* Physical disability (non-ambulatory patient e.g. wheelchair or bed-bound)
* Inability to obtain informed consent
* Cognitive failure making them unable to give consent or understand questionnaires or instruction.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with known Pulmonary Sarcoidosis according to ATS/ERS/ WASOG criteria statement ascertained by self-reporting.
Sampling Method: Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2017-11-07 (Actual); Primary Completion 2018-06-15 (Actual); Study Completion 2018-06-15 (Actual)

PRIMARY OUTCOMES:
Daily physical activity measures against self-reported by tri-axial accelerometry | 7 days
  minutes of physical activity per day

SECONDARY OUTCOMES:
Functional exercise capacity | 14 days
  Six-minute walk test (Distance in meters)
Muscle strength (isokinetic dynamometer) | 14 days
  Peak torque (Nm)
Lung function using spirometry | 14 days
  Lung volume (L/min)
Quality of Life Score | 14 days
  Patient reported health status using Sarcoidosis Health Questionnaire score
Body Composition | 1 day
  Body pat percentage (BF %)
Anthropometric weight | 1 day
  Body mass (kg)
Anthropometric height | 1 day
  body stature (cm)
Cardiovascular Health | 14 days
  Blood pressure (mmHg)
Cardiovascular function | 14 days
  Heart rate (bpm)
Oxygen saturation | 14 days
  SaP02 %
Borg rate of perceived exertion | 14 days
  RPE scale (6-20)
Borg Dyspnoea | 14 days
  Scale (0-10)
Fatigue Assessment Scale | 14 days
  Likert scale (1-5)

CONTACTS AND LOCATIONS:
Overall Officials: Juliet Parry, Study Chair — Kingston University
Locations (2):
- United Kingdom (2):
  - Applied & Human Sciences Human Performance Lab, Kingston upon Thames, Surrey
  - Kingston University London, Kingston upon Thames, Surrey

IPD SHARING:
Plan to Share IPD: Undecided
The results of the study will form part of the researcher's Masters (MSc) by Research thesis and may be published anonymously in professional journals and/or as conference presentations.

REFERENCES:
- [Background] Strookappe B, Saketkoo LA, Elfferich M, Holland A, De Vries J, Knevel T, Drent M. Physical activity and training in sarcoidosis: review and experience-based recommendations. Expert Rev Respir Med. 2016 Oct;10(10):1057-68. doi: 10.1080/17476348.2016.1227244. Epub 2016 Sep 8. PMID 27552344
- [Background] Holland AE, Dowman LM, Hill CJ. Principles of rehabilitation and reactivation: interstitial lung disease, sarcoidosis and rheumatoid disease with respiratory involvement. Respiration. 2015;89(2):89-99. doi: 10.1159/000370126. Epub 2015 Jan 21. PMID 25633076
- [Background] Judson MA, Chaudhry H, Louis A, Lee K, Yucel R. The effect of corticosteroids on quality of life in a sarcoidosis clinic: the results of a propensity analysis. Respir Med. 2015 Apr;109(4):526-31. doi: 10.1016/j.rmed.2015.01.019. Epub 2015 Feb 7. PMID 25698652
- [Background] Alhamad EH, Shaik SA, Idrees MM, Alanezi MO, Isnani AC. Outcome measures of the 6 minute walk test: relationships with physiologic and computed tomography findings in patients with sarcoidosis. BMC Pulm Med. 2010 Aug 9;10:42. doi: 10.1186/1471-2466-10-42. PMID 20696064
- [Background] Karadalli MN, Bosnak-Guclu M, Camcioglu B, Kokturk N, Turktas H. Effects of Inspiratory Muscle Training in Subjects With Sarcoidosis: A Randomized Controlled Clinical Trial. Respir Care. 2016 Apr;61(4):483-94. doi: 10.4187/respcare.04312. Epub 2015 Dec 29. PMID 26715771
- [Background] Huppmann P, Sczepanski B, Boensch M, Winterkamp S, Schonheit-Kenn U, Neurohr C, Behr J, Kenn K. Effects of inpatient pulmonary rehabilitation in patients with interstitial lung disease. Eur Respir J. 2013 Aug;42(2):444-53. doi: 10.1183/09031936.00081512. Epub 2012 Oct 25. PMID 23100507
- [Background] Cox CE, Donohue JF, Brown CD, Kataria YP, Judson MA. The Sarcoidosis Health Questionnaire: a new measure of health-related quality of life. Am J Respir Crit Care Med. 2003 Aug 1;168(3):323-9. doi: 10.1164/rccm.200211-1343OC. Epub 2003 May 8. PMID 12738606
- [Background] De Vries J, Michielsen H, Van Heck GL, Drent M. Measuring fatigue in sarcoidosis: the Fatigue Assessment Scale (FAS). Br J Health Psychol. 2004 Sep;9(Pt 3):279-91. doi: 10.1348/1359107041557048. PMID 15296678
- [Background] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- [Background] Butland RJ, Pang J, Gross ER, Woodcock AA, Geddes DM. Two-, six-, and 12-minute walking tests in respiratory disease. Br Med J (Clin Res Ed). 1982 May 29;284(6329):1607-8. doi: 10.1136/bmj.284.6329.1607. No abstract available. PMID 6805625
- [Background] Parcell AC, Sawyer RD, Tricoli VA, Chinevere TD. Minimum rest period for strength recovery during a common isokinetic testing protocol. Med Sci Sports Exerc. 2002 Jun;34(6):1018-22. doi: 10.1097/00005768-200206000-00018. PMID 12048331

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-11-07): https://cdn.clinicaltrials.gov/large-docs/36/NCT03336736/Prot_SAP_002.pdf
  • Informed Consent Form (2017-11-07): https://cdn.clinicaltrials.gov/large-docs/36/NCT03336736/ICF_003.pdf